CLINICAL TRIAL: NCT01605318
Title: A Phase I/II Study of Once or Twice Weekly IMMU-130 (hMN-14-SN38, Antibody-Drug Conjugate) in Patients With Colorectal Cancer
Brief Title: Study of Labetuzumab Govitecan in Participants With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMMU-130-02
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Colorectal Cancer; Colon Cancer; Rectal Cancer
Keywords: Previously treated Metastatic colorectal cancer; Previously treated Colon cancer; Previously treated Rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — labetuzumab govitecan; Immunoconjugates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase1: Dose-escalation Phase: Labetuzumab Govitecan (LG) Once Weekly Dosing (Experimental): Participants will receive 8, 12 and 16 mg/dose of LG once weekly dosing until unacceptable toxicity, progressive disease or death whichever occurs first, for each 21-day cycle for up to up to 8 cycles, with a contingency to examine intermediate dose levels of 10 or 14 mg/kg, or if necessary to a lower dose level of 6 mg/kg.
  Interventions: Drug: Labetuzumab Govitecan (LG)
- Phase1: Dose-escalation Phase: LG Twice Weekly Dosing (Experimental): Participants will receive 6 and 9 mg/kg per dose twice weekly dose of LG until unacceptable toxicity, progressive disease or death whichever occurs first, for each 21-day cycle for up to up to 8 cycles. A lower dose level of 4 mg/kg may be added if > 1 out of 3 or 2 out of 6 participants are unable to tolerate all 4 doses without dose delay or reduction.
  Interventions: Drug: Labetuzumab Govitecan (LG)
- Phase 2: Dose-expansion Phase: LG Once or Twice Weekly Dosing (Experimental): Participants will receive selected doses of LG once or twice weekly until unacceptable toxicity, progressive disease or death whichever occurs first, for each 21-day cycle for up to 8 cycles.
  Interventions: Drug: Labetuzumab Govitecan (LG)

INTERVENTIONS:
Drug: Labetuzumab Govitecan (LG) — Administered as a slow intravenous (IV) infusion.
  Other Names: hMN14-SN38; Labetuzumab-SN38; Antibody-Drug Conjugate; IMMU-0130; GS-0130

SUMMARY:
The goal of this clinical study is to determine the dosing and safety of labetuzumab govitecan (formerly known as IMMU-130; hMN-14-SN38, antibody-drug conjugate) in participants with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed colorectal adenocarcinoma.
* Stage IV (metastatic) disease.
* Previously treated with at least one prior irinotecan-containing regimen for colorectal cancer.
* Adequate performance status (Eastern Cooperative Oncology Group (ECOG) 0 or 1).
* Expected survival > 6 months.
* Carcinoembryonic antigen (CEA) plasma levels > 5 ng/mL.
* Measurable disease by computed tomography (CT) or Magnetic resonance imaging (MRI).
* At least 4 weeks beyond treatment (chemotherapy, immunotherapy and/or radiation therapy) or major surgery and recovered from all acute toxicities.
* At least 2 weeks beyond corticosteroids.
* Adequate hematology without ongoing transfusional support (hemoglobin > 9 g/dL, absolute neutrophil count (ANC) > 1,500 per mm^3, platelets > 100,000 per mm^3).
* Adequate renal and hepatic function (creatinine ≤ 1.5 x IULN, bilirubin ≤ institutional upper limit of normal (IULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x IULN or 5 x IULN if know liver metastases).
* Otherwise, all toxicity at study entry ≤ Grade 1 by National cancer institute common terminology criteria for adverse events (NCI CTC) v4.0.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Women of childbearing potential and fertile men unwilling to use effective contraception during study until conclusion of 12-week post-treatment evaluation period.
* Individuals with Gilbert's disease or known central nervous system (CNS) metastatic disease.
* Individuals with CEA plasma levels > 1000 ng/mL must be approved in advance by the Sponsor.
* Presence of bulky disease (defined as any single mass > 10 cm in its greatest dimension).
* Individuals with active ≥ grade 2 anorexia, nausea or vomiting, and/or signs of intestinal obstruction.
* Individuals with non-melanoma skin cancer or carcinoma in situ of the cervix are eligible, while individuals with other prior malignancies must have had at least a 3-year disease-free interval.
* Individuals known to be human immunodeficiency virus (HIV) positive, hepatitis B positive, or hepatitis C positive.
* Known history of unstable angina, myocardial infarction, or congestive heart failure present within 6 months or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy.
* Known history of clinically significant active chronic obstructive pulmonary disease (COPD), or other moderate-to-severe chronic respiratory illness present within 6 months.
* Infection requiring intravenous antibiotic use within 1 week.
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-02-12 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events and Serious Adverse Events (SAEs) | From first dose date up to approximately 2 years after the last dose or until disease progression
Percentage of Participants With Laboratory Abnormalities | From first dose date up to approximately 2 years after the last dose or until disease progression

SECONDARY OUTCOMES:
Duration of Response | From first documentation of PR or CR to the earlier of the first documentation of PD or death from any cause (Up to approximately 2 years after the last dose or until disease progression)
  Duration of response (DOR) is defined as the interval from the first documentation of PR or CR to the earlier of the first documentation of disease progression (PD) or death from any cause.
Progression-free Survival | From first dose date up to 12 weeks post treatment (Up to approximately 2 years after the last dose or until disease progression)
  Progression free survival (PFS) is defined as the interval from the start of study drug treatment to the earlier of the first documentation of disease progression or death from any cause.
Time to Progression | From first dose of study treatment up to PD (Up to approximately 2 years after the last dose or until disease progression)
  Time to progression is defined as the interval from the first dose of treatment to the first documentation of disease progression (PD).
Overall Survival | From first dose date up to approximately 2 years
  Overall survival is defined as the time from start of study drug treatment to death from any cause.
Time-to-treatment Failure | From first dose date up to 8 treatment cycles (each cycle = 21 days) (Up to approximately 24 weeks)
  Time to treatment failure (TTF) is defined as the interval from the start of treatment to the earlier of the first documentation of disease progression or death due to any cause, the permanent cessation of LG therapy due to all reasons except progressive disease, participant died or lost to follow up.
Change from Baseline in Carcinoembryonic Antigen (CEA) Serum Levels | From first dose date up to approximately 2 years after the last dose or until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (7):
- United States (7):
  - UCLA Jonsson Comprehensive Cancer Center, Santa Monica, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Helen F. Graham Cancer Center-Christiana Care, Newark, Delaware
  - IUHealth Goshen Center for Cancer Care, Goshen, Indiana
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fox Chase, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Govindan SV, Goldenberg DM. New antibody conjugates in cancer therapy. ScientificWorldJournal. 2010 Oct 12;10:2070-89. doi: 10.1100/tsw.2010.191. PMID 20953556
- [Background] Govindan SV, Cardillo TM, Moon SJ, Hansen HJ, Goldenberg DM. CEACAM5-targeted therapy of human colonic and pancreatic cancer xenografts with potent labetuzumab-SN-38 immunoconjugates. Clin Cancer Res. 2009 Oct 1;15(19):6052-61. doi: 10.1158/1078-0432.CCR-09-0586. Epub 2009 Sep 29. PMID 19789330
- [Background] Moon SJ, Govindan SV, Cardillo TM, D'Souza CA, Hansen HJ, Goldenberg DM. Antibody conjugates of 7-ethyl-10-hydroxycamptothecin (SN-38) for targeted cancer chemotherapy. J Med Chem. 2008 Nov 13;51(21):6916-26. doi: 10.1021/jm800719t. Epub 2008 Oct 22. PMID 18939816
- [Background] Govindan SV, Griffiths GL, Hansen HJ, Horak ID, Goldenberg DM. Cancer therapy with radiolabeled and drug/toxin-conjugated antibodies. Technol Cancer Res Treat. 2005 Aug;4(4):375-91. doi: 10.1177/153303460500400406. PMID 16029057
- [Background] Dotan E, Cohen SJ, Starodub AN, Lieu CH, Messersmith WA, Simpson PS, Guarino MJ, Marshall JL, Goldberg RM, Hecht JR, Wegener WA, Sharkey RM, Govindan SV, Goldenberg DM, Berlin JD. Phase I/II Trial of Labetuzumab Govitecan (Anti-CEACAM5/SN-38 Antibody-Drug Conjugate) in Patients With Refractory or Relapsing Metastatic Colorectal Cancer. J Clin Oncol. 2017 Oct 10;35(29):3338-3346. doi: 10.1200/JCO.2017.73.9011. Epub 2017 Aug 17. PMID 28817371